CLINICAL TRIAL: NCT04848948
Title: Effects of Short-term Calory Restriction and Biofeedback on Anthropometric and Metabolic Parameters as Well as Biological and Psychological Stress Correlates in Healthy Women
Brief Title: Impact of Calory Restriction and Biofeedback on Endocrine and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Prof.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-GI-01
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Neuroendocrinology; Mental Stress; Psychological; Obesity
MeSH Terms: conditions — Stress, Psychological; Obesity | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- F.X.Mayr & Biofeedback (Experimental): two weeks of F.X. Mayr diet and biofeedback
  Interventions: Behavioral: Calory Restriction (F.X. Mayr & VLCD); Behavioral: Biofeedback
- F.X.Mayr (Active Comparator): two weeks of F.X. Mayr diet
  Interventions: Behavioral: Calory Restriction (F.X. Mayr & VLCD)
- VLCD & Biofeedback (Experimental): two weeks of very low calorie diet and biofeedback
  Interventions: Behavioral: Calory Restriction (F.X. Mayr & VLCD); Behavioral: Biofeedback
- VLCD (Active Comparator): two weeks of very low calorie diet
  Interventions: Behavioral: Calory Restriction (F.X. Mayr & VLCD)

INTERVENTIONS:
Behavioral: Calory Restriction (F.X. Mayr & VLCD) — VLCD restricts calory intake to 630 - 700 kcal per day (20% fat, 34% protein, 46% carbohydrates).
  F.X. Mayr diet similarly applies calorie restriction to 700 - 800 kcal per day and includes daily ingestion of isotonic magnesium sulfate solution.
Behavioral: Biofeedback — Three sessions of biofeedback (50 minutes) over a time frame of 14 days, aimed at improving biological functions and especially heart-rate-variability under stress condition.
  Arms: F.X.Mayr & Biofeedback; VLCD & Biofeedback

SUMMARY:
Backgroup/relevance: Overweight and obesity, defined by a respective body mass index of above 25 and 30 kg/m2, are getting increasingly common in all regions of the world. Obesity is currently estimated to be present in more than 10% of the global population while overweight roughly reached an estimate of 40% in 2016.

Overweight dramatically increases the risk for a wide range of disorders such as diabetes mellitus and other metabolic and cardiovascular disorders subsumed under the term metabolic syndrome, increasing the risk for life-threatening cardiovascular events such as myocardial infarction and stroke. Similar to other chronic diseases such as mental health disorders, prescribing medication was oftentimes insufficient and should be complemented by patient empowerment to reach sufficient treatment adherence and control of lifestyle factors. Thereby, overweight and obesity can easily be challenged by patients themselves without pharmacological intervention.

Overweight may place central in the crossroad between metabolic and mental health for several reasons. Excessive body fat is known to cause subclinical inflammation that was also associated with many psychiatric disorders such as major depression. Similarly, the hypothalamic-pituitary-adrenal axis relevant for stress response was shown to be dysregulated in both metabolic and mental health disorders.

Study design: In this study, non-pharmacological interventions are applied in healthy women with overweight or obesity and self-perceived psychological stress. Women staying at the "la pura" women´s health resort (www.lapura.at/) are invited to partake in the study and receive a short-term intervention of calory restriction. Thereby, either F.X. Mayr or very-low-calory-diet (VLCD) will be applied, reducing calory intake to 700-800 kcal/die. Following random assigment to four treatment arms, half of the women also receive a 7-session clinical-psychological intervention consisting of biofeedback, individualized psycho-education on stress prevention and mindlessness training.

Women are assessed at baseline and after two weeks of interventions for metabolic parameters such as insulin functioning, anthropometric parameters such as body weight and body fat, blood parameters such as sex hormones, fat metabolism and liver function, parameters of neuroplasticity such as brain derived neurotrophic factor (BDNF), as well as psychological and biological stress correlates and mental health symptom dimensions.

ELIGIBILITY:
Inclusion Criteria:

* women willing to undergo two-weeks of calory restriction
* at least 18 years of age

Exclusion Criteria:

* currently pregnant
* any acute or a severe chronic illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
PSS score | Baseline, changes over two weeks
  Perceived Stress Scale total score
BODI | Baseline, changes over two weeks
  buron-out-diagnostic-inventory scores, 4 summary items and 3 stress self-ratings
BSI | Baseline, changes over two weeks
  Brief Symptom Inventory, 9 dimensional subscores and global severity score
waist-to-height ratio | Baseline
  Anthropometric parameter
HbA1c | Baseline
  Glycated hemoglobin
HOMA-IR | Baseline
  Functional parameter for insulin resistance
Matsuda Index | Baseline
  Functional parameter for insulin sensitivity
Body mass index | Baseline, changes over two weeks
  weight in relation to height
HRV | Baseline, changes over two weeks
  heart rate variability

SECONDARY OUTCOMES:
Body fat | Baseline, changes over two weeks
  measured by bioimpedance analysis
lean mass | Baseline, changes over two weeks
  measured by bioimpedance analysis
Phase angle | Baseline, changes over two weeks
  ratio of reactance versus electric resistance, measured by bioimpedance analysis
Resistin | Baseline, changes over two weeks
  Adipocines
Leptin | Baseline, changes over two weeks
  Adipocines
Secretagogin | Baseline, changes over two weeks
  Adipocines
Adiponectin | Baseline, changes over two weeks
  Adipocines
BDNF | Baseline, changes over two weeks
  brain derived neurotrophic factor
Estrogen | Baseline, changes over two weeks
  Sex hormone
Testosterone | Baseline, changes over two weeks
  Sex hormone
Luteinizing hormone | Baseline, changes over two weeks
  Sex hormone
Follicle-stimulating hormone | Baseline, changes over two weeks
  Sex hormone
Total cholesterol | Baseline, changes over two weeks
  Lipid metabolism
High-density lipoprotein (HDL) | Baseline, changes over two weeks
  Lipid metabolism
BSRI | Baseline
  Bem sex role inventory, female, male, neutral scores

CONTACTS AND LOCATIONS:
Locations (1):
- VAMED Gender Insitute, Gars am Kamp, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Upon request